CLINICAL TRIAL: NCT03309670
Title: Psychiatric Future of Young Patients Hospitalized in the Pass'Aje Service Between 2006 and 2010
Acronym: After Pass'Aje
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-355
Record Dates: First submitted 2017-10-02; First posted 2017-10-13 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Psychiatry
Keywords: psychiatric outcome; psychosocial outcome; young

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Formers young patients: all patients hospitalized between 2006 and 2010 in the Pass'Aje unit
  Interventions: Other: Psychiatric future

INTERVENTIONS:
Other: Psychiatric future — Former young psychiatric patients are contacted to determine their psychiatric outcome.

SUMMARY:
The emergence of adult psychic disorders occurs in about three quarters of cases before 25 years. The Pass-Aje service of Clermont-Ferrand University Hospital is a psychiatric unit specializing in the management of disorders of young adults. This unit evaluates the first episodes among the diversity of the clinical presentations of the psychic disorders. Suicidal attempts or ideations account for a large part of the reasons for entering the unit and are found transversely in many disorders. Among the reasons for hospitalization are a wide variety of situations that are not initially associated with an accurate diagnosis such as withdrawal, de-schooling, runaways, behavioral disorders (disorders of social interactions, self and hetero aggression, eating disorders).

Investigator propose to study the psychiatric outcome of hospitalized patients in the Pass-Aje unit and their psychosocial evolution in order to compare them with the data of the general population and to identify the factors influencing their future.

DETAILED DESCRIPTION:
Former young psychiatric patients hospitalized in the Pass'Aje units are contacted by phone several years later to determine their psychiatric outcome.

ELIGIBILITY:
Inclusion Criteria:

* all patients hospitalized in the Pass'Aje unit between 2006 and 2010
* Aged from 16 to 25 years when hospitalized

Exclusion Criteria:

* Patient refusing or not understanding the purpose of the study.
* Patients who died.
* Patient phone number unavailable or non-functional

Ages: 23 Years to 36 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young patients hospitalized in psychiatric service
Sampling Method: Non-Probability Sample
Enrollment: 660 (Estimated)
Dates: Start 2017-09-14 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2019-05-15 (Estimated)

PRIMARY OUTCOMES:
Psychiatric rehospitalisation | at day 1 during the phone call
  the psychiatric outcome comprises 3 parameters :
  * ongoing psychiatric follow-up (yes / no)
  * psychotropic treatment in progress (yes / no)
  * psychiatric hospitalizations after the first hospitalization in Pass'Aje (yes / no)

SECONDARY OUTCOMES:
Determination of social outcomes | at day 1 during the phone call
  Educational level of obtained by patients will be compared to data of the general population according to sex, age and parents' social environment
Percentage of patients with an occupational activity | at day 1 during the phone call
  Percentage of patients with an occupational activity will be compared to data of the general population according to sex, age and parents' social environment

CONTACTS AND LOCATIONS:
Overall Officials: Eve COURTY, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France